CLINICAL TRIAL: NCT01398137
Title: An Observational Multi-Centre Field Study to Assess Symptom Scores and Rescue Medication Usage in Subjects With a History of Ragweed Allergen-Induced Rhinoconjunctivitis
Brief Title: Ragweed Observational Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TR003
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Ragweed Allergy
Keywords: Ragweed allergy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ragweed allergic subjects

SUMMARY:
This is an observational to evaluate Total Rhinoconjunctivitis Symptom Score and rescue medication usage (as measured by Rescue Medication Score as a Combined Score to inform the design of a phase III field study with ToleroMune Ragweed.

ELIGIBILITY:
Inclusion Criteria

* Male or female, aged 18-65 years.
* Reliable history of rhinoconjunctivitis and/or rhinoconjunctivitis plus controlled asthma on exposure to ragweed allergen for at least 2 years and required symptomatic treatment for at least 1 year.
* Positive skin prick test (SPT) to Ambrosia artemisiifolia
* Specific Immunoglobulin E (IgE) against Ambrosia artemisiifolia >0.35 kU/L

Exclusion Criteria

* Positive skin test to any confounding, co-existing seasonal allergens likely to be present during the Pre-season baseline and ragweed pollen periods (grasses, miscellaneous weeds, fall trees) and who have received medication for these confounding seasonal allergies.
* Medical records of symptomatic perennial allergic rhinitis and/or asthma due to an allergen to which the subject is regularly exposed (moulds, dust mites, cockroaches, and animal dander) and have received medication for these perennial allergies
* Subjects with a history of severe drug allergy, severe angioedema or anaphylactic reaction to food or previous SPT for any allergen.
* Subjects with a history of any significant disease or disorder (e.g., cardiovascular, pulmonary, gastrointestinal, liver, renal, neurological, immunopathological, musculoskeletal, endocrine, metabolic, malignant, psychiatric, major physical impairment) which, in the opinion of the Investigator, may influence the subject's ability to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a history of ragweed allergy for at least 2 years and which required symptomatic treatment for at least 1 year
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Mean daily Combined Score during the site-specific ragweed pollen period | Daily during ragweed season expected to last approximately 8 weeks
  Combined score is the Total Rhinoconjunctivitis Score(TRSS)/8 added to the Rescue Medication Score

SECONDARY OUTCOMES:
Mean Combined Score during the site-specific peak ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean TRSS during the site-specific ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean TRSS during the site-specific peak ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean Rescue Medication Score during the site-specific ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean Rescue Medication Score during the site-specific peak ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean component scores of the TRSS (nasal and non nasal) during the site specific ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean component scores of the TRSS (nasal and non nasal) during the site specific peak ragweed pollen period | Through 2011 ragweed season expected to last approximately 8 weeks
Mean Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) score during the site specific peak ragweed pollen period in a subset of the study population | Through 2011 ragweed season approximately 8 weeks
Weeks of partly controlled or uncontrolled asthma | Through 2011 ragweed season expected to last approximately 8 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Owensboro, Kentucky
  - Minneapolis, Minnesota
  - Plymouth, Minnesota
  - Rolla, Missouri
  - St Louis, Missouri
  - Warrensburg, Missouri
  - High Point, North Carolina
  - Canton, Ohio
  - Springfield, Virginia
  - Greenfield, Wisconsin